CLINICAL TRIAL: NCT00785642
Title: Safety Dermatological Evaluation: Genital Mucous Irritation - Product Tested: Dermacyd PH_DETINLYN Tangerine Mix (Lactic Acid).
Brief Title: Dermacyd PH_DETINLYN Tangerine Mix (Lactic Acid) - Safety.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04304
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Dermacyd PH_DETINLYN Tangerine Mix (Lactic Acid)
  Interventions: Drug: Dermacyd PH_DETINLYN Tangerine Mix (Lactic Acid)

INTERVENTIONS:
Drug: Dermacyd PH_DETINLYN Tangerine Mix (Lactic Acid)

SUMMARY:
To prove the safety of the gynaecological formulation in normal conditions of use.

ELIGIBILITY:
Inclusion criteria:

* Integral skin test in the region;
* Use of cosmetic product of the same category;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time;

Exclusion criteria:

* Lactation or gestational risk or gestation;
* Use of Anti-inflammatory, immunosuppression or antihistaminic drugs;
* Atopic antecedent or allergic to cosmetic product;
* Active cutaneous disease in the evaluation area;
* Diseases which cause immunology decrease, such as diabetes and HIV;
* Endocrinal pathologies;
* Intense solar exposure 15 days before the evaluation;
* Treatment until four months before the selection

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 10 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The absence of irritation and the good acceptability will be evaluated using one specific scale which describes the intensity of the reaction. | From the treatment start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil